CLINICAL TRIAL: NCT06280313
Title: Impact of Splenectomy on the Efficacy of Targeted Therapy and Immunotherapy in Unresectable HCC Patients With Cirrhotic Portal Hypertension
Status: Recruiting | Type: Observational
Sponsor: Zhiyong Huang (Other)
Collaborators: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); Zhongnan Hospital (Other); Renmin Hospital of Wuhan University (Other); Taihe Hospital (Other); Hubei Cancer Hospital (Other); Xiangyang Central Hospital (Other); Wuhan Central Hospital (Other); Yichang Third Renmin Hospital (Unknown)
Responsible Party: Sponsor-Investigator, Zhiyong Huang, Professor, Tongji Hospital
Organization: Tongji Hospital (Other)
Other Study IDs: uHCC-STI-TJ01
Record Dates: First submitted 2024-02-20; First posted 2024-02-28 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Unresectable Hepatocellular Carcinoma
Keywords: Immunotherapy; Targeted therapy; Splenectomy; HCC

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Treatment (Splenectomy+Targeted therapy+ Immunotherapy): Eligible patients with unresectable hepatocellular carcinoma accompanied by cirrhotic portal hypertension were enrolled in the trial, and all participants underwent either open or laparoscopic splenectomy, with or without devascularization around the cardia. Starting two weeks post-surgery, patients began intravenous infusion of PD-1 monoclonal antibody, Tislelizumab, at a dosage of 200mg every three weeks. Three weeks post-surgery, patients commenced oral administration of the targeted therapy, Lenvatinib, with a dosage based on body weight: 8mg (≤60kg) or 12mg (>60kg), once daily.
  Interventions: Combination Product: Splenectomy+Targeted therapy+ Immunotherapy

INTERVENTIONS:
Combination Product: Splenectomy+Targeted therapy+ Immunotherapy — Eligible patients with unresectable hepatocellular carcinoma accompanied by cirrhotic portal hypertension were enrolled in the trial, and all participants underwent either open or laparoscopic splenectomy, with or without devascularization around the cardia. Starting two weeks post-surgery, patients began intravenous infusion of PD-1 monoclonal antibody, Tislelizumab, at a dosage of 200mg every three weeks. Three weeks post-surgery, patients commenced oral administration of the targeted therapy, Lenvatinib, with a dosage based on body weight: 8mg (≤60kg) or 12mg (>60kg), once daily.

SUMMARY:
Currently, the combination of targeted therapy and immunotherapy is the first-line treatment for advanced hepatocellular carcinoma (HCC). However, a subset of HCC patients with severe splenomegaly, splenic hyperfunction, and esophagogastric varices due to liver cirrhosis and portal hypertension may be unable to undergo or sustain the combination therapy, ultimately missing the optimal treatment window. Prior studies have indicated that splenectomy can significantly improve liver function and hepatic reserve in cirrhotic patients. It also addresses splenic hyperfunction and reduces the risk of bleeding from esophagogastric varices by combining splenectomy with devascularization around the cardia. Additionally, splenectomy contributes to the improvement of liver fibrosis and restoration of immune function in cirrhotic patients. This study aims to elucidate the impact of splenectomy on the efficacy of combination targeted and immunotherapy in unresectable HCC patients with cirrhotic portal hypertension, particularly those with poor liver function, significant splenic hyperfunction, and severe esophagogastric varices. The research also seeks to explore whether changes in the tumor immune microenvironment before and after splenectomy can influence the effectiveness of immunotherapy. Ultimately, the goal is to provide therapeutic opportunities for this specific patient population.

DETAILED DESCRIPTION:
This is a single-arm, open-label, observational study assessing the impact of splenectomy on the efficacy of combined targeted and immune therapy in patients with unresectable hepatocellular carcinoma accompanied by cirrhotic portal hypertension. Eligible patients with unresectable hepatocellular carcinoma were enrolled in the trial, and all participants underwent either open or laparoscopic splenectomy, with or without devascularization around the cardia. Starting two weeks post-surgery, patients began intravenous infusion of PD-1 monoclonal antibody, Tislelizumab, at a dosage of 200mg every three weeks. Three weeks post-surgery, patients commenced oral administration of the targeted therapy, Lenvatinib, with a dosage based on body weight: 8mg (≤60kg) or 12mg (>60kg), once daily. The use of Tislelizumab and Lenvatinib continued until the primary endpoint, which was disease progression, intolerable toxicity reactions, or other criteria specified in the protocol for terminating the study treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18 to 75 years (inclusive).
2. No prior systemic antitumor treatment or meeting the criteria for splenectomy during treatment.
3. Clinical or pathological diagnosis of hepatocellular carcinoma (HCC) that is unresectable initially or has recurred after surgery.
4. HBV-DNA less than 1*10^5 copies/ml and undergoing antiviral therapy.
5. ECOG performance status score of 0-1, without significant organ dysfunction.
6. Child-Pugh score of 5-7.
7. Spleen thickness >4.0 cm.
8. History of esophagogastric varices, red signs, or variceal bleeding with or without splenomegaly.
9. Splenomegaly with WBC <2.5 × 10^9/L and PLT <70 × 10^9/L, or splenomegaly with WBC <2.0 × 10^9/L or PLT <50 × 10^9/L.
10. Important organ functions meeting the following criteria: Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3*ULN, total bilirubin ≤ 3*ULN; International normalized ratio (INR) ≤ 1.5*ULN; prothrombin time ≤ 1.5*ULN; creatinine ≤ 1.5*ULN.
11. Able to undergo local treatments such as transarterial chemoembolization (TACE), hepatic artery infusion chemotherapy (HAIC), selective internal radiation therapy with yttrium-90 (SIRT), stereotactic body radiation therapy (SBRT), and ablation (including radiofrequency ablation (RFA) and microwave ablation (MWA)).
12. Willing to provide informed consent.
13. Expected survival time of more than 3 months.

Exclusion Criteria:

1. History of or concurrent active malignancy (excluding malignancies that have been cured for over 5 years or in situ cancers that can be completely cured with adequate treatment).
2. Presence of central nervous system metastasis or a history of brain metastasis.
3. History of organ transplantation.
4. History of surgery in the head, chest, or abdomen within the past six months.
5. Child-Pugh class C liver function or significant ascites.
6. Marked thrombosis in the portal venous system or extensive cancer thrombus in the main portal vein.
7. Activated partial thromboplastin time (APTT) or prothrombin time (PT) exceeding 1.5 times the upper limit of normal (as per the normal values of the clinical trial research center), or evidence of bleeding tendency or history of bleeding within the two months prior to enrollment, regardless of severity.
8. Ongoing active infection within 7 days after completion of systemic antibiotic therapy.
9. Active coronary artery disease, severe/unstable angina, or newly diagnosed angina or myocardial infarction within the past 12 months before enrollment.
10. Thrombotic or embolic events within the past 12 months, such as cerebrovascular accidents (including transient ischemic attacks), pulmonary embolism, or deep vein thrombosis.
11. New York Heart Association (NYHA) class II or above congestive heart failure.
12. Human immunodeficiency virus (HIV) infection or known acquired immunodeficiency syndrome (AIDS), positive syphilis serology, untreated active hepatitis (defined as HBV-DNA ≥ 10^5 copies/ml; HCV-RNA higher than the lower limit of detection for the assay).
13. Any active, known, or suspected autoimmune disease. Stable subjects not requiring systemic immunosuppressive therapy may be included, such as those with type 1 diabetes, hypothyroidism requiring only hormone replacement therapy, and skin diseases not requiring systemic treatment (e.g., vitiligo, psoriasis, and alopecia).
14. Interstitial lung disease, non-infectious pneumonia, or uncontrolled systemic diseases (e.g., diabetes, hypertension, pulmonary fibrosis, and acute pneumonia).
15. Pregnant or lactating women or females with a positive pregnancy test prior to the first dose who have the potential for pregnancy.
16. The investigator deems the subject inappropriate for participation in this clinical study due to any clinical or laboratory abnormalities or compliance issues.
17. Severe psychological or mental abnormalities.
18. Participation in another drug clinical trial within the past 4 weeks.
19. Other reasons that the investigator considers unsuitable for enrollment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Unresectable HCC patients with cirrhotic portal hypertension
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-03-15 (Actual); Primary Completion 2027-03-15 (Estimated); Study Completion 2028-03-15 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | 6 weeks after first dose of Tislelizumab
  ORR refers to the proportion of patients whose tumors shrink to a certain amount and maintain for a certain period of time (6 weeks after first dose of Tislelizumab), including CR+PR cases. CR (complete remission): disappearance of all target lesions, PR (partial remission): reduction of the sum of the length and diameter of the baseline lesions by ≥30%

SECONDARY OUTCOMES:
Overall Survival (OS) | through study completion, an average of 2 year
  OS was defined as time from diagnosis to death from any cause or the last follow-up
Progression Free Survival (PFS) | 18 months
  PFS refers to the time from subject enrollment to disease progression according the Response Evaluation Criteria in Solid Tumors version 1.1 (RECISTv1.1) or death

CONTACTS AND LOCATIONS:
Overall Officials: Zhiyong Huang, Principal Investigator — Tongji Hospital
Locations (1):
- Tongji Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No